CLINICAL TRIAL: NCT00682435
Title: Safety and Speed of Onsent of Intravenous Hydromorphone Using Incremental 1mg Doses up to 2mg in the Treatment of Adult ED Patients With Moderate to Severe Pain
Brief Title: Safety Study of Intravenous Hydromorphone Using Incremental 1mg Doses up to 2mg for Adult ED Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, MD, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC0702028
Record Dates: First submitted 2008-05-19; First posted 2008-05-22 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: Nonelderly patients with acute moderate to severe pain
MeSH Terms: conditions — Pain | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydromorphone (Experimental): 1 mg IV hydromorphone, + optional 1 mg IV hydromorphone 15 minutes later
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — 1mg IV hydromorphone, followed by an optional dose of 1mg IV hydromorphone 15 minutes later if the patient answers "yes" to the question, "Do you want more pain medication?"
  Other Names: Dilaudid

SUMMARY:
We wish to examine the safety and speed of onset of giving a dose of 1mg hydromorphone followed by an additional 1mg. Eligible patients will be given 1 mg intravenous (IV) hydromorphone. At 15 minutes, these patients will be asked the question, "Do you need more pain medication?" Those that answer "yes" will receive an additional 1mg IV hydromorphone. Those that answer "no" will not receive additional pain medications at that time period (15 minutes). Thus, we wish to give up to 2 mg IV hydromorphone titrated to patients' pain, which we believe will result in less incidence of oxygen desaturation.

If our study shows that this regimen is safe, its efficacy can be assessed in future trials. Positive results of those trials may lead to the use of this regimen to improve pain management in the emergency department.

DETAILED DESCRIPTION:
Prospective interventional study at an urban academic emergency department (ED). One milligram of IV hydromorphone was administered to adults 21 to 64 years of age who had acute severe pain. Fifteen minutes later, patients were asked whether they wanted more pain medication. If they answered yes, they received another 1 mg of IV hydromorphone and were again asked 15 minutes later whether they wanted more pain medication. The primary efficacy outcome was the proportion of patients who had adequate analgesia, defined as declining additional hydromorphone within 1 hour of entering the protocol. The primary safety outcome was incidence of oxygen desaturation less than 95%. Secondary outcomes included numeric rating scale pain scores and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 21 years: Patients under the age of 21 are automatically triaged to the Children's Hospital at Montefiore Emergency Department, and hence cannot be enrolled in this study.
2. Age less than 65 years of age: Patients age 65 and over will be excluded in this study as the effects on opioids on the elderly may be different than in the non-elderly.
3. Pain with onset within 7 days: Pain within seven days is the definition of acute pain that has been used in ED literature.
4. ED attending physician's judgment that patient's pain warrants use of morphine: The factors that influence the decision to use parenteral opioids are complex and extensive. An approach that is commonly taken to address the issue of patient selection in drug trials is to use a specific condition (e.g., renal colic) or treatment (e.g., post-hysterectomy) that would generally be thought to be appropriately treated with an opioid analgesic, thereby eliminating individual judgment about eligibility for the study. However in order to assess the role of hydromorphone with the widest generalizability in the ED setting, we decided to enroll patients with a variety of diagnoses, all with a complaint of acute pain. Opioids are not an appropriate treatment for all patients who present with a complaint of pain (e.g., gastroenteritis, migraine). Therefore, unless there is a restriction to patients with a specific diagnosis, either a comprehensive list of diagnoses and situations in which opioids are indicated must be specified, or clinical judgment needs to be used. We have opted for the latter alternative.
5. The use of patients with a variety of diagnoses, and therefore heterogeneous painful stimuli, risks masking a treatment effect because of large inter-individual variability. There are several design and analytic factors (detailed below) that attenuate this risk: 1) a sufficiently large number of patients will be randomly assigned to each group so that the variety of painful stimuli will be equally distributed between treatment groups; 2) change in pain intensity and pain relief will be analyzed rather than absolute pain intensity or pain relief therefore reducing variability.
6. Normal mental status: In order to provide measures of pain experienced the patient needs to have a normal mental status. Orientation to person, place and time will be used as an indicator of sufficiently normal mental status to participate in the study.

Exclusion Criteria:

1. Prior use of methadone: the effect of methadone use on the perception of acute pain is unknown and suspected to be altered. We feel that the needs of patients on methadone may exceed the dosage ceiling of 2mg that will be used for this study. Similar to sickle cell patients and chronic cancer patients, patients on methadone usually require significantly higher doses of opioids to control their pain. Thus, we feel that it would be unethical to restrict the dose that this subset of patients can receive.
2. Use of other opioids or tramadol within past seven days: to avoid introducing bias related to opioid tolerance that may alter the response to the study medication thereby masking the medication's effect.
3. Prior adverse reaction to hydromorphone.
4. Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months result in alteration in pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, migraine, and peripheral neuropathies.
5. Alcohol intoxication: the presence of alcohol intoxication as judged by the treating physician may alter perception, report, and treatment of pain.
6. Systolic Blood Pressure <90 mm Hg: Hydromorphone can produce peripheral vasodilation that may result in orthostatic hypotension or syncope.
7. Oxygen saturation <95% on room air: For this study, oxygen saturation must be 95% or above on room air in order to be enrolled.
8. Use of monoamine oxidase (MAO) inhibitors in past 30 days: MAOs have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant respiratory depression or coma.
9. C02 measurement greater than 46: In accordance with a similar study (04-12-360), three subsets of patients will have their CO2 measured using a handheld capnometer prior to enrollment in the study. If the CO2 measurement is greater than 46, then the patient will be excluded from the study. The 3 subsets are as follows:

   1. All patients who have a history of chronic obstructive pulmonary disease (COPD)
   2. All patients who report a history of asthma together with greater than a 20 pack-year smoking history
   3. All patients reporting less than a 20 pack-year smoking history who are having an asthma exacerbation
10. Pregnancy: this will be determined by asking the female of reproductive age about her pregnancy status and/or through the results of urine or serum pregnancy test.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chang, M.D., Principal Investigator — Motefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydromorphone
Started | 230
Ensured Enrolled Only Once | 228
Sufficient Data to Carry Out Analysis | 223
Completed | 223
Not Completed | 7
Not completed — Insufficient data | 5
Not completed — Erroneously enrolled twice | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hydromorphone
Number analyzed (Participants) | 223
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [30 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144
  Male | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 134
  Black | 65
  White | 15
  Other | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 223
Weight [Median (Inter-Quartile Range); unit: lbs] | 179 [147 to 200]
Location of pain [Count of Participants; unit: Participants]
  Abdomen | 149
  Other | 74
Pain intensity [Count of Participants; unit: Participants] — Pain intensity is measured on the numerical rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable)
  Participants
    4-6 | 12
    7 | 17
    8 | 39
    9 | 36
    10 | 119
Number of participants experiencing Nausea or Vomiting before baseline [Count of Participants; unit: Participants]
  Yes | 85
  No | 138

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had Adequate Analgesia
Description: Adequate analgesia is defined as declining additional hydromorphone within 1 hour of entering the protocol
Time Frame: 60 minutes after medication infused
Population: Those given a second dose only included patients who wanted more pain medication 15 minutes after 1st dose. 7 patients did not receive the second dose, resulting in 44 patients analyzed instead of expected 51
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 223
Participants
  15 minutes after 1st 1mg dose of IV hydromorphone: wanted more pain medication | 51
  15 minutes after 1st 1mg dose of IV hydromorphone: Did not want more pain medication | 172
  15 minutes after 2nd 1 mg dose of IV hydromorphone: number analyzed (Participants) | 44
  15 minutes after 2nd 1 mg dose of IV hydromorphone: wanted more pain medication | 9
  15 minutes after 2nd 1 mg dose of IV hydromorphone: Did not want more pain medication | 35

2. Primary Outcome: Number of Patients With Oxygen Desaturation Less Than 95%
Description: primary safety outcome, defined as number of participants who experienced oxygen saturation < 95%
Time Frame: 120 minutes after medication infused
Population: Total of 223 split into patients who received only 1 mg of IV hydromorphone (179) and those who received 2 mg of IV hydromorphone
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 223
Participants
  1 mg IV hydromorphone: number analyzed (Participants) | 179
  1 mg IV hydromorphone | 11
  2 mg IV hydromorphone: number analyzed (Participants) | 44
  2 mg IV hydromorphone | 0

3. Secondary Outcome: Number of Patients With Reduction in Pain Intensity
Description: Pain intensity is measured on the numerical rating scale (NRS), with a pain score from 0 (no pain) to 10 (worst pain imaginable). The reduction in pain intensity is defined here as a change in pain score by 2 or more units.
Time Frame: 60 minutes after medication infused
Measure: Number; unit: % of participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 223
% of participants | 86

4. Secondary Outcome: Change in Pain Intensity
Description: Pain intensity is measured on the numerical rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable) from baseline to 60 minutes after medication infused
Time Frame: 60 minutes after medication infused
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 223
units on a scale | 6 [4 to 8]

ADVERSE EVENTS:
Time Frame: 60 minutes
Groups:
- 1 mg Hydromorphone: 1 mg IV hydromorphone, + optional 1 mg IV hydromorphone 15 minutes later
  Hydromorphone: 1mg IV hydromorphone, followed by an optional dose of 1mg IV hydromorphone 15 minutes later if the patient answers "yes" to the question, "Do you want more pain medication?"
Arm/Group | 1 mg Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/223
Serious Adverse Events (participants affected / at risk) | 0/223
Other Adverse Events (participants affected / at risk) | 83/223
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 1 mg Hydromorphone (N=223)
Oxygen saturation < 95% (Respiratory, thoracic and mediastinal disorders) | 11
Pulse rate < 60 beats/min (Cardiac disorders) | 21/219 — excludes patients with baseline pulse rate less than 60 beats/min
Systolic blood pressure < 100 mmHg (Vascular disorders) | 2
Respiratory rate < 12 breaths/min (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 25/138 — excludes patients who were nauseated or vomiting before administration of first 1 mg of IV hydromorphone
Vomiting (Gastrointestinal disorders) | 9/138 — excludes patients who were nauseated or vomiting before administration of first 1 mg IV hydromorphone
Pruritus (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes